CLINICAL TRIAL: NCT06009133
Title: Surgical Excision Versus Medical Treatment in Acute External Thrombosed Hemorrhoidal Disease
Brief Title: Surgical Approach for Acute External Thrombosed Hemorrhoidal Disease
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Principle Investigator, Konya Meram State Hospital
Other Study IDs: Konya HH Group
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhoids External Thrombosed
MeSH Terms: interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative Treatment Group: Micronized purified flavonoid fraction, which is routinely used within indications in hemorrhoidal disease and recommended in ESCP and ASCRS guidelines, and licensed for use in hemorrhoidal disease by the Ministry of Health in our country, was given 2 g/day for one month.
  Also, Conservative methods (fiber foods, warm shower, regulation of toilet habits, laxatives and nonsteroidal anti-inflammatory drugs) were recommended.
  Interventions: Procedure: Conservative treatment
- Surgical Treatment Group: While the patient was in the Jack-knife position, both hips were pulled laterally with tapes, appropriate visualization was obtained, the external thrombosed pack was excised under local anesthesia, and the wound was left to heal with secondary intention.Conservative methods were recommended in the surgical group as well as in the medical group.
  Interventions: Procedure: Surgical Treatment

INTERVENTIONS:
Procedure: Conservative treatment — Micronized purified flavonoid fraction, which is routinely used within indications in hemorrhoidal disease and recommended in ESCP and ASCRS guidelines, and licensed for use in hemorrhoidal disease by the Ministry of Health in our country, was given 2 g/day for one month.
  Also, Conservative methods (fiber foods, warm shower, regulation of toilet habits, laxatives and nonsteroidal anti-inflammatory drugs) were recommended.
  Groups: Conservative Treatment Group
Procedure: Surgical Treatment — While the patient was in the Jack-knife position, both hips were pulled laterally with tapes, appropriate visualization was obtained, the external thrombosed pack was excised under local anesthesia, and the wound was left to heal with secondary intention.Conservative methods were recommended in the surgical group as well as in the medical group.
  Groups: Surgical Treatment Group

SUMMARY:
Acute external thrombosed hemorrhoidal disease (AETHH) is one of the emergent complications of hemorrhoidal disease that results in pain and loss of work force. Although surgical excision is recommended in the treatment of AETHH in the guidelines of the American Society of Colorectal Surgeons (ASCRS) and the European Society of Coloproctology (ESCP), the level of evidence is low and it is emphasized that additional studies are needed. Therefore, the investigators aimed to compare the efficacy of surgical excision with medical treatment in the treatment of AETHH.

DETAILED DESCRIPTION:
Hemorrhoids are normal anatomical structures and are divided into internal and external according to the dentate line. External hemorrhoids distal to the dentate line, unlike internal hemorrhoids, are covered with squamous epithelium (anoderm), have somatic innervation, and are highly sensitive to pain.

While internal hemorrhoidal disease causes symptoms such as painless bleeding, mucosal prolapse, soiling, and itching, external hemorrhoids do not cause clinical findings unless thrombosed. Acute constipation or excessive straining are held responsible for acute external thrombosed hemorrhoidal disease (AETHD). It appears as a painful, firm, purple-colored mass in the anoderm, and the main symptom is anal pain. The severity of pain increases in the first 24-48 hours after the formation of the thrombosed pack and reaches its peak. The pain is quite severe in the first 72-96 hours. Afterwards, with the resorption of the thrombosis, the severity of the pain decreases and the disease heals, leaving a skin tag behind.

AETHD can be treated with surgical excision or conservative approaches. Conservative treatment includes a warm water sitz bath, analgesics, anti-inflammatory drugs. Also, phlebotonic drugs can be added. In the ASCRS and ESCP guidelines, early surgical excision is recommended for patients with acute external thrombosed hemorrhoidal disease in the first 72-96 hours (low quality evidence 2C). Guidelines highlight the lack of controlled studies of AETHD treatment .

In this study, the investigators aimed to compare early surgical excision with conservative treatment in terms of pain control and recurrence in the treatment of AETHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-70 who present with isolated external thrombosed hemorrhoids
* Patients with the onset of the complaint before 96 hours

Exclusion Criteria:

Patients under the age of 18 and patients over the age of 70

* Mentally retarded patients
* Pregnant patients
* Patients with concomitant proctological disorders (anal fissure, anal fistula, anal abscess, etc.)

Those with a history of proctology surgery

* Patients with grade 3-4 internal hemorrhoids
* Patients using anticoagulant drugs
* Patients whose complaint has passed 96 hours after onset

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of patients who applied to the general surgery outpatient clinic due to acute external thrombosed hemorrhoids disease. Patients who fully met the inclusion criteria and did not meet the exclusion criteria constituted the sample group.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Pain score with visual analog scale | 12 hours
  The participants pain at the 12th hour postoperatively was scored with a visual analog scale. The visual analog scale was between 0 and 10 mm. 0 rated as no pain, 10 as very severe pain.

SECONDARY OUTCOMES:
Time to return to daily activities | 15 days
  The patients' return to daily activities were recorded.
Recurrence | 6 months
  It was recorded whether the patients had hemorrhoid recurrence at 6 months.
Satisfaction survey | 6 months
  The satisfaction level of the participants was scored on a visual analog scale six months after the treatment. The visual analog scale was between 0 and 10 mm. 0 was rated as not at all satisfied, and 10 was rated as very satisfied.
  Satisfaction questionnaire was applied to the patients at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Yaldız, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)